CLINICAL TRIAL: NCT05339165
Title: FAMily Factors INvolved in Eating Disorders
Acronym: FamFINED
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Thomas Meyer, Head of Laboratory, University Medical Center Goettingen
Other Study IDs: 32/1/17
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Eating Disorders
Keywords: Eating disorder, anorexia nervosa, bulimia nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Psychotherapy

SUMMARY:
This observational study compares parental age and birth order in patients diagnosed with anorexia nervosa and bulimia nervosa.

DETAILED DESCRIPTION:
Study participants are recruited (300 patients for each entity). Healthy subjects without evidence of an eating disorder serve as a control group. Psychometric assessment will include data on pathological eating behavior and general psychological and interpersonal problems.

Outcome measures The SCL-90-R questionnaire is a self-report inventory for adolescents and adults that assesses a wide range of psychological problems and symptoms of psychopathology. The questionnaire consists of 90 items, each of which contributes to one of nine primary symptom dimensions.

The short form of the Inventory of Interpersonal Problems (IIP-C) is used to measure interpersonal problems. This self-report questionnaire contains 64 items assigned to eight subscales.

Eligible candidates are stratified as cases or matched controls as follows:

1. Cases are eligible patients diagnosed with anorexia nervosa or bulimia nervosa (n=300 for each entity) at the time of study inclusion.
2. Controls (100) are healthy subjects of a similar age distribution and from the same study site without the diagnosis of an eating disorder.

Inclusion criteria:

- Age > 12 and < 59 years (adolescents and adults).

Exclusion criteria:

* Diagnosed with a malignant disease
* Not fluent in the German language
* Severe mental disorder

ELIGIBILITY:
Inclusion Criteria:

- Age > 12 and < 59 years (adolescents and adults) with either anorexia nervosa or bulimia nervosa.

Exclusion Criteria:

* Diagnosed with a malignant disease
* Not fluent in the German language
* Severe mental disorder

Ages: 12 Years to 59 Years | Sex: All
Age Groups: Child, Adult
Study Population: Study participants with diagnosed anorexia nervosa or bulimia nervosa according to ICD-10 criteria
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
SCL-90-R questionnaire | One day
  The SCL-90-R questionnaire is a self-report inventory for adolescents and adults that assesses a wide range of psychological problems and symptoms of psychopathology. The questionnaire consists of 90 items, each of which contributes to one of nine primary symptom dimensions.
Short form of the Inventory of Interpersonal Problems (IIP-C) | One day
  The short form of the Inventory of Interpersonal Problems (IIP-C) is used to measure interpersonal problems. This self-report questionnaire contains 64 items assigned to eight subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, Principal Investigator — University of Göttingen
Locations (2):
- Germany (2):
  - University of Göttingen, Göttingen, NDS
  - University Medical Center, Göttingen

IPD SHARING:
Plan to Share IPD: No